CLINICAL TRIAL: NCT00610272
Title: Investigation of Optimal Radiotherapy Regimen and Type of Irradiation in Treatment of Painful Bone Metastasis
Brief Title: Optimization of Radiotherapy in Treatment of Painful Bone Metastasis
Acronym: bone mets
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E33028
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Pain; Bone Metastasis
Keywords: single bone metastasis; multiple bone metastasis; pain relief; radiotherapy
MeSH Terms: conditions — Pain | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Single Site Radiation 4Gy Fraction (Experimental): 4 Gy single fraction; mandate first retreatment if moderate or severe pain persists or recurs (as measured by categorical pain scale or VAS greater than 50 mm), >4 weeks after initial RT) retreat with 8 Gy single fraction; second retreatment is optional if moderate or severe pain recurs (as measured by categorical pain scale or VAS greater than 50 mm), retreat with 8 Gy after > 4 weeks
  Interventions: Radiation: Radiotherapy
- Single Site Radiation 8Gy Fraction (Active Comparator): 8 Gy single fraction, mandate first retreatment if moderate or severe pain persists or recurs (as measured by categorical pain scale or VAS greater than 50 mm), >4 weeks after initial RT) retreat with 8 Gy single fraction; second retreatment is optional if moderate or severe pain recurs (as measured by categorical pain scale or VAS greater than 50 mm), retreat with 8 Gy after > 4 weeks
  Interventions: Radiation: Radiotherapy
- Multiple Sites Radiation 8Gy Fraction (Active Comparator): 8 Gy in a single fraction; retreatments > 4 weeks, using local RT fields to sites of residual or recurrent, moderate or severe pain with a single fraction of 8 Gy) ; second reirradiation with 8 Gy using local RT fields optional (at discretion of PI);
  Interventions: Radiation: Radiotherapy
- Multiple Sites Radiation 12Gy Fraction (Experimental): 12 Gy in 4 fractions of 3 Gy in 2 consecutive days interfraction interval of a minimum of 6 hrs; retreatments > 4 weeks using local RT fields to sites of residual or recurrent, moderate or severe pain with a single fraction of 8 Gy); second reirradiation with 8 Gy using local RT fields optional (at discretion of PI) ;
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — 4 Gy single fraction; mandate first retreatment if moderate or severe pain persists or recurs (as measured by categorical pain scale or VAS greater than 50 mm), >4 weeks after initial RT) retreat with 8 Gy single fraction; second retreatment is optional if moderate or severe pain recurs (as measured by categorical pain scale or VAS greater than 50 mm), retreat with 8 Gy after > 4 weeks
  Arms: Single Site Radiation 4Gy Fraction
Radiation: Radiotherapy — 8 Gy single fraction, mandate first retreatment if moderate or severe pain persists or recurs (as measured by categorical pain scale or VAS greater than 50 mm), >4 weeks after initial RT) retreat with 8 Gy single fraction; second retreatment is optional if moderate or severe pain recurs (as measured by categorical pain scale or VAS greater than 50 mm), retreat with 8 Gy after > 4 weeks
  Arms: Single Site Radiation 8Gy Fraction
Radiation: Radiotherapy — 8 Gy in a single fraction; retreatments > 4 weeks, using local RT fields to sites of residual or recurrent, moderate or severe pain with a single fraction of 8 Gy) ; second reirradiation with 8 Gy using local RT fields optional (at discretion of PI);
  Arms: Multiple Sites Radiation 8Gy Fraction
Radiation: Radiotherapy — 12 Gy in 4 fractions of 3 Gy in 2 consecutive days interfraction interval of a minimum of 6 hrs; retreatments > 4 weeks using local RT fields to sites of residual or recurrent, moderate or severe pain with a single fraction of 8 Gy); second reirradiation with 8 Gy using local RT fields optional (at discretion of PI) ;
  Arms: Multiple Sites Radiation 12Gy Fraction

SUMMARY:
Bone metastasis is one of the most frequent end complications of the cancer. Radiation therapy is the mainstay of treatment in this disease. Single fraction radiotherapy in both single and multiple bone metastasis is widely used, but optimization of the single dose fractionation is needed. Two different regimens of radiotherapy dose fractionation will be investigated in both single and multiple bone metastasis and endpoints will include pain relief as well as toxicity and quality of life.

DETAILED DESCRIPTION:
PROTOCOL SCHEMA

Group A Treatment of single site of painful bone metastasis:

Arm 1: 4 Gy single fraction; mandate first retreatment if moderate or severe pain persists or recurs (as measured by categorical pain scale or VAS greater than 50 mm), >4 weeks after initial RT) retreat with 8 Gy single fraction; second retreatment is optional if moderate or severe pain recurs (as measured by categorical pain scale or VAS greater than 50 mm), retreat with 8 Gy after > 4 weeks

Arm 2: 8 Gy single fraction, mandate first retreatment if moderate or severe pain persists or recurs (as measured by categorical pain scale or VAS greater than 50 mm), >4 weeks after initial RT) retreat with 8 Gy single fraction; second retreatment is optional if moderate or severe pain recurs (as measured by categorical pain scale or VAS greater than 50 mm), retreat with 8 Gy after > 4 weeks

Group B Treatment of multiple bone metastasis: lower hemibody radiotherapy (LHBI):

Arm 3: 8 Gy in a single fraction; retreatments > 4 weeks, using local RT fields to sites of residual or recurrent, moderate or severe pain with a single fraction of 8 Gy) ; second reirradiation with 8 Gy using local RT fields optional (at discretion of PI);

Arm 4: 12 Gy in 4 fractions of 3 Gy in 2 consecutive days interfraction interval of a minimum of 6 hrs; retreatments > 4 weeks using local RT fields to sites of residual or recurrent, moderate or severe pain with a single fraction of 8 Gy); second reirradiation with 8 Gy using local RT fields optional (at discretion of PI) ;

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of malignancy associated with radiological evidence of painful bone metastasis
* If patients with two sites of pain requiring separate treatment are to be entered, the same randomized treatment option will be used for both sites, but response at each site will be scored and analyzed separately.
* age > 18 years
* anticipated remaining life of at least 12 weeks (3 months)
* informed consent

Exclusion Criteria:

* Primary histology myeloma
* Sites of previous RT or previous radioisotope treatment
* conditions or circumstances, which may interfere with treatment or follow-up
* complicated bone metastasis (pathological fractures, metastatic spinal cord compression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2008-01; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Pain Relief (response rate) at 4 weeks | Up to 52 weeks

SECONDARY OUTCOMES:
Onset and Duration of Pain Relief in Responders | Up to 52 weeks
Toxicity | Up to 52 weeks
Quality of Life | Up to 52 weeks
Rates of Pathological Fractures and Spinal Cord Compression | Up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elena Fidarova, MD, Study Chair — International Atomic Energy Agency
Locations (12):
- Centre Pierre et Marie Curie, Centre hospitalier universitaire Mustapha (CHU), Algiers, Algeria
- Irmandade de Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Brazil
- Misr Oncology Center (MOC), Cairo, Egypt
- Tata Memorial Hospital, Mumbai, India
- Institute of Oncology, University of Vilinius, Vilnius, Lithuania
- Instituto Nacional de Cancerología (INCAN), Mexico City, Mexico
- Institute of Radiotherapy and Oncology, Skopje, North Macedonia
- Institute of Oncology and Radiology, Belgrade, Serbia
- Spain (2):
  - Hospital Clinic Universidad de Barcelona, Barcelona
  - Hospital Son Dureta, Palma de Mallorca
- Institut national de cancer Salah Azaiz, Tunis, Tunisia
- Mount Vernon Cancer Centre, Northwood, United Kingdom

REFERENCES:
- [Background] Salazar OM, DaMotta NW, Bridgman SM, Cardiges NM, Slawson RG. Fractionated half-body irradiation for pain palliation in widely metastatic cancers: comparison with single dose. Int J Radiat Oncol Biol Phys. 1996 Aug 1;36(1):49-60. doi: 10.1016/s0360-3016(96)00248-9. PMID 8823258
- [Background] Salazar OM, Sandhu T, da Motta NW, Escutia MA, Lanzos-Gonzales E, Mouelle-Sone A, Moscol A, Zaharia M, Zaman S. Fractionated half-body irradiation (HBI) for the rapid palliation of widespread, symptomatic, metastatic bone disease: a randomized Phase III trial of the International Atomic Energy Agency (IAEA). Int J Radiat Oncol Biol Phys. 2001 Jul 1;50(3):765-75. doi: 10.1016/s0360-3016(01)01495-x. PMID 11395246
- [Background] Mithal NP, Needham PR, Hoskin PJ. Retreatment with radiotherapy for painful bone metastases. Int J Radiat Oncol Biol Phys. 1994 Jul 30;29(5):1011-4. doi: 10.1016/0360-3016(94)90396-4. PMID 7521863
- [Background] Hoskin PJ, Price P, Easton D, Regan J, Austin D, Palmer S, Yarnold JR. A prospective randomised trial of 4 Gy or 8 Gy single doses in the treatment of metastatic bone pain. Radiother Oncol. 1992 Feb;23(2):74-8. doi: 10.1016/0167-8140(92)90338-u. PMID 1372126
- [Background] Wu JS, Wong R, Johnston M, Bezjak A, Whelan T; Cancer Care Ontario Practice Guidelines Initiative Supportive Care Group. Meta-analysis of dose-fractionation radiotherapy trials for the palliation of painful bone metastases. Int J Radiat Oncol Biol Phys. 2003 Mar 1;55(3):594-605. doi: 10.1016/s0360-3016(02)04147-0. PMID 12573746
- [Background] Gaze MN, Kelly CG, Kerr GR, Cull A, Cowie VJ, Gregor A, Howard GC, Rodger A. Pain relief and quality of life following radiotherapy for bone metastases: a randomised trial of two fractionation schedules. Radiother Oncol. 1997 Nov;45(2):109-16. doi: 10.1016/s0167-8140(97)00101-1. PMID 9423999
- [Background] Arcangeli G, Micheli A, Arcangeli G, Giannarelli D, La Pasta O, Tollis A, Vitullo A, Ghera S, Benassi M. The responsiveness of bone metastases to radiotherapy: the effect of site, histology and radiation dose on pain relief. Radiother Oncol. 1989 Feb;14(2):95-101. doi: 10.1016/0167-8140(89)90053-4. PMID 2469105